CLINICAL TRIAL: NCT00353184
Title: Randomized Controlled Trial of Oral Montelukast Added to Standard Therapy for Acute Asthma Exacerbations in Children Age 6 to 14 Years
Brief Title: Montelukast Added to Standard Therapy for Acute Asthma in Children Age 6-14 Years
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results of the interim analysis suggested no significant diff between study groups.
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Academy of Pediatrics (Other); Ambulatory Pediatric Association (Other)
Responsible Party: Kyle Nelson, Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WUSM HSC #01-0464
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Asthma
Keywords: Acute; Asthma; Child; Pediatric; Emergency; Oral; Montelukast; Forced Expiratory Volume in One Second; FEV1
MeSH Terms: conditions — Asthma; Emergencies | interventions — montelukast

INTERVENTIONS:
Drug: Montelukast 5-mg orally added to standard therapy

SUMMARY:
Oral montelukast is helpful in chronic asthma. The purpose of this pediatric study was to investigate whether the addition of oral montelukast to standard therapy for acute asthma exacerbations results in further improvement in breathing function over three hours.

DETAILED DESCRIPTION:
We hypothesized that children with moderate acute asthma exacerbations receiving oral montelukast in addition to standard therapy will have at least 12% greater FEV1 improvement in three hours than those receiving standard therapy alone.

In this randomized double-blind placebo-controlled study, we enrolled emergency patients aged 6-14 years with moderate acute asthma exacerbations (initial PEFR 40-70% predicted). Subjects received montelukast 5-mg or placebo orally then standard therapy consisting of weight-based doses of nebulized albuterol, nebulized ipratropium bromide, and oral corticosteroids. We measured FEV1 before study medication administration and hourly for three hours.

We conducted a planned an interim analysis after approximately one-half of the estimated sample had been enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Seeking care in ED for acute asthma exacerbation
* Age 6-14 years inclusive
* Initial FEV1 = 40-70% predicted (defined as moderate severity)
* Consent to participate in study

Exclusion Criteria:

* Severe exacerbation requiring immediate therapy as determined by treating clinician
* Pregnancy by history
* Cystic Fibrosis by history
* Tuberculosis
* Gastroesophageal reflux disease requiring medications
* Acute or chronic liver disease
* Bronchopulmonary dysplasia
* Premature <34 weeks gestational age by history
* Having used leukotriene-modifying medication within 48 hours
* Having used theophylline within four weeks
* Unable to perform FEV1

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2001-09; Primary Completion 2004-10 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in One Second (FEV1)

SECONDARY OUTCOMES:
Hospitalization Rate
Relapse Visit Rate

CONTACTS AND LOCATIONS:
Overall Officials: Kyle A Nelson, MD, Principal Investigator — Physician in Division of Pediatric Emergency Medicine at Washington University School of Medicine in St. Louis; David M Jaffe, MD, Study Chair — Senior Advisor for Study, Division Director for Pediatric Emergency Medicine at Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States